CLINICAL TRIAL: NCT02348320
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of a Personalized Polyepitope DNA Vaccine Strategy in Breast Cancer Patients With Persistent Triple-Negative Disease Following Neoadjuvant Chemotherapy
Brief Title: Safety and Immunogenicity of a Personalized Polyepitope DNA Vaccine Strategy in Breast Cancer Patients With Persistent Triple-Negative Disease Following Neoadjuvant Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201505074
Record Dates: First submitted 2015-01-21; First posted 2015-01-28 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2019-06

CONDITIONS: Triple Negative Breast Cancer; Triple-Negative Breast Cancer; Triple Negative Breast Neoplasms
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Personalized polyepitope DNA vaccine (Experimental): Participants will be treated by electroporation with 4 mg of a personalized polyepitope DNA vaccine at Day 1, Day 29 (+/1- 7 days), and Day 57 (+/- 7 days) with at least 21 days between injection days. Each DNA vaccination with be 4 mg vaccine administered intramuscularly using a TriGrid electroporation device.
  Interventions: Biological: Personalized polyepitope DNA vaccine

INTERVENTIONS:
Biological: Personalized polyepitope DNA vaccine

SUMMARY:
This is a phase 1 open-label study to evaluate the safety and immunogenicity of a personalized polyepitope DNA vaccine strategy. The personalized polyepitope DNA vaccines will be formulated as naked plasmid DNA vaccines. The hypothesis of this study is that personalized polyepitope DNA vaccines will be safe for human administration and capable of generating measurable CD8 T cell responses to mutant tumor-specific antigens.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of invasive breast cancer.
* ER and PR less than Allred score of 3 or less than 1% positive staining cells in the invasive component of the tumor. Patients not meeting this pathology criteria, but have been clinically treated as having TNBC, can be enrolled at PI discretion.
* HER2 negative by FISH or IHC staining 0 or 1+.
* Consented for genome sequencing and dbGAP-based data sharing and has provided or will provide germline and tumor DNA samples of adequate quality for sequencing. Fresh tissue is preferred (from biopsy at the time of port placement) but archival tissue is allowed
* Clinical stage T1c-T4c, any N, M0 primary tumor by AJCC 7th edition clinical staging prior to neoadjuvant chemotherapy, with residual invasive breast cancer after neoadjuvant therapy. If the patient has invasive cancer in the contralateral breast, she is not eligible for this study.
* At least 18 years of age. Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Adequate organ and marrow function no more than 14 days prior to registration as defined below:

  * WBC ≥ 3,000/μL
  * absolute neutrophil count ≥1,500/μL
  * platelets ≥ 100,000/μL
  * total bilirubin ≤ 2.5 X institutional upper limit of normal
  * AST/ALT ≤ 2.5 X institutional upper limit of normal
  * creatinine ≤ 1.5 X institutional upper limit of normal
* Women of reproductive potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Evidence of progressive breast cancer within the last 30 days.
* Received chemotherapy, radiotherapy, or biologic therapy within the last 30 days (neoadjuvant chemotherapy excluded).
* Experiencing any clinically significant adverse events above Grade 1 (according to CTCAE 4.0) due to agents administered more than 30 days earlier. However, patients with Grade 2 Alopecia will be considered eligible.
* Receiving any other investigational agent(s) or has received an investigational agent within the last 30 days.
* Known metastatic disease.
* Invasive cancer in the contralateral breast.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (including sinus bradycardia), or psychiatric illness/social situation that would limit compliance with study requirements.
* Prior or currently active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines. Asthma or chronic obstructive pulmonary disease that does not require daily systemic corticosteroids is acceptable. Any patients receiving steroids should be discussed with the PI to determine if eligible.
* Pregnant or breastfeeding. A negative serum pregnancy test is required no more than 7 days before study entry.
* The patient with a previous history of non-breast malignancy is eligible for this study only if the patient meets the following criteria for a cancer survivor. A cancer survivor is eligible provided the following criteria are met: (1) patient has undergone potentially curative therapy for all prior malignancies, (2) patients have been considered disease free for at least 1 year (with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix).
* Patient must have no active major medical or psychosocial problems that could be complicated by study participation.
* Known HIV-positive status. These patients are ineligible because of the potential inability to generate an immune response to vaccines.
* Subjects with a strong likelihood of non-adherence such as difficulties in adhering to follow-up schedule due to geographic distance from the Siteman Cancer Center should not knowingly be registered.
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for eligible injection sites (left and right medial deltoid region) exceeds 40 mm.
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art.
* Therapeutic or traumatic metal implant in the skin or muscle of either deltoid region.
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical examination, EKG, and/or laboratory screening test
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child
* Syncopal episode within 12 months of screening
* Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06-17 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Safety of the personalized polyepitope DNA vaccine strategy, measured by both clinical observation and laboratory evaluation | 52 weeks
  Assessment of plasmid DNA safety will include both clinical observation and laboratory evaluation. Safety will be closely monitored after injection with eight or more clinical and laboratory assessments in the first 24 weeks of the trial. The following parameters will be assessed following vaccination:
  1. Local signs and symptoms
  2. Systemic signs and symptoms
  3. Laboratory evaluations, including blood counts and serum chemistries
  4. Adverse, and serious adverse events

SECONDARY OUTCOMES:
Immunogenicity of the personalized polyepitope DNA vaccine strategy, measured by ELISPOT analysis, a surrogate for CD8 T cell function, and multiparametric flow cytometry | 52 weeks
  Immunogenicity will be measured by ELISPOT analysis, a surrogate for CD8 T cell function, and multiparametric flow cytometry. In both assays the quantity and quality of antigen-specific CD8 T cells is determined; the ELISPOT analysis is based on measuring the frequencies of IFN-γ producing T cells in response to polyepitope antigen, whereas the multiparametric flow cytometry assesses phenotypic as well as functional characteristics of epitope-specific CD8 T cells. In the proposed study, blood samples will be collected at multiple time points (n=8) and PBMC isolated and cryopreserved. Upon completion of the vaccination protocol, all samples will be analyzed simultaneously in order to minimize assay-to-assay variation.

CONTACTS AND LOCATIONS:
Overall Officials: William E Gillanders, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Goedegebuure SP, Chen MY, Mishra R, Zhang F, Yu YY, Singhal K, Li L, Gao F, Myers NB, Vickery T, Hundal J, McLellan MD, Sturmoski MA, Kim SW, Chen I, Davidson JT 4th, Sankpal NV, Myles S, Suresh R, Ma CX, Foluso A, Wang-Gillam A, Davies S, Hagemann IS, Mardis ER, Griffith O, Griffith M, Miller CA, Hansen TH, Fleming TP, Schreiber RD, Gillanders WE. Neoantigen DNA vaccines are safe, feasible, and induce neoantigen-specific immune responses in triple-negative breast cancer patients. Genome Med. 2024 Nov 14;16(1):131. doi: 10.1186/s13073-024-01388-3. PMID 39538331
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu